CLINICAL TRIAL: NCT06379191
Title: The Efficacy of WeChat-based Multidisciplinary Full-course Nutritional Management Program on the Nutritional Status of Ovarian Cancer Patients Undergoing Chemotherapy: a Randomized Controlled Trial
Brief Title: The Efficacy of WeChat-based Multidisciplinary Full-course Nutritional Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZS-3411
Record Dates: First submitted 2024-02-25; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Cancer
Keywords: WeChat; nutrition management; ovarian cancer; chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care group (Placebo Comparator): Upon admission, patients were provided with admission counselling, explained the complications associated with chemotherapy, and given a chemotherapy care booklet and a leaflet on diet and nutrition. Before discharge, the patients were given the nutritional guidebook again. Responsible nurses made one telephone follow-up visit between chemotherapy sessions.
  Interventions: Behavioral: Nutrition intervention model based on WeChat applets
- Intervention group (Experimental): Patients were instructed to search for the "Good Nutrition" applet on WeChat and added it to their "My Applets" for easy access. The patient was informed of the users' nameand password. The patient was introduced to the main functional sections of the applet and the content settings of each section to become familiar with the applet. Patients were invited to join our nutrition management group chat. At the same time, patients were allowed to choose to have a private chat with a member of the nutrition management team via WeChat at any time.
  Interventions: Behavioral: Nutrition intervention model based on WeChat applets

INTERVENTIONS:
Behavioral: Nutrition intervention model based on WeChat applets — We recorded the full nutritional management plan for ovarian cancer chemotherapy patients obtained through evidence-based in the previous period into the applet developed by our team - "Good Nutrition". At the first chemotherapy admission assessment, patients were instructed to search for the applet on WeChat and add it to "My applet". The patient was introduced to the main functional sections of the applet and the content settings for each section. The patient was instructed to turn on the applet notification permission and set it to receive new content alerts. Patients were invited to join our nutrition management group chat. They were informed that throughout the intervention phase, we would be sending evidence-based scientific articles to the group chat for independent study, and that they were allowed to ask questions, share personal experiences, and discuss lifestyles within the group.

SUMMARY:
As the most malignant type of cancer in the female reproductive system, ovarian cancer (OC) has become the second leading cause of death among Chinese women. Chemotherapy is the main treatment for OC patients, and its numerous adverse effects can easily lead to malnutrition. It is difficult to centrally manage OC patients in the intervals between chemotherapy. The utility of WeChat, an effective and more cost-efficient mobile tool, in chronic disease management has been highlighted.

DETAILED DESCRIPTION:
Ovarian cancer (OC) is the most malignant type of tumor in the female reproductive system with poor prognosis. According to the latest statistics, there are 196,000 estimated OC cases, 45,000 estimated new cases, and 29,000 estimated OC deaths in China, making this disease become the second leading cause of death among Chinese women.

Approximately 90% of patients with OC receive chemotherapy. The carboplatin-paclitaxel combination as a first-line chemotherapy regimen for OC has shown considerable efficacy over the past 30 years. Unfortunately, one of the major adverse effects of chemotherapy is malnutrition. Malnutrition is defined as a nutritional condition in which deficiencies of energy, protein and other nutrients have measurable adverse effects on tissue/body form, function and clinical outcomes. The most common adverse effects of chemotherapy, including anorexia, altered taste and smell, food aversions, nausea and vomiting, mucositis, xerostomia, constipation, diarrhea and early satiety, negatively affect nutritional status. Malnutrition has been shown to be one of the leading causes of death in OC patients. It not only severely diminishes the efficacy of treatment, but leads to increased complications, decreased quality of life, prolonged hospitalization, increased healthcare costs, and shorter survival time. However, existing nutritional interventions lack personalized guidance for patients' nutritional status and symptoms during chemotherapy. In addition, it is difficult to centrally manage patients who are homebound between chemotherapy. Therefore, the construction of personalized nutritional management programs and the development of innovative telemedicine interventions for OC patients undergoing chemotherapy has become an urgent issue.

WeChat, a very popular social application in China, has more than 1 billion monthly active users. It is easy to operate and offers multiple functions such as text and voice messaging, free voice and video calls, group chats, subscription to public accounts and applets, etc. WeChat has been demonstrated to be an effective and more cost-efficient technological tool for chronic disease management. Currently, the application of WeChat in cancer patients mainly focuses on discharge follow-up, symptom management, cancer prevention, and intervention of psychological problems. The effect of WeChat application in nutritional management of cancer patients has not been explored. Therefore, the aim of this study was to implement a continuous follow-up strategy and health monitoring based on a WeChat platform for OC patients undergoing chemotherapy during the chemotherapy interval to ensure that each phase of chemotherapy is delivered on schedule and to improve the survival rate of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

≥18 years

Pathologically confirmed ovarian cancer

Paclitaxel combined with carboplatin as a chemotherapy regimen

Normal cognitive ability and proficiency in the use of WeChat

Exclusion Criteria:

Malignant tumor of another system

Serious illness or failure of vital organs such as the heart, lungs, liver and kidneys

Receiving enteral or parenteral nutritional support

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
patient-generated subjective global assessment (PG-SGA) | T0=before the first admission to the hospital for chemotherapy, T1=2 weeks after the first chemotherapy, and T6=2 weeks after the sixth chemotherapy
  PG-SGA was used as a prognostic tool developed specifically for patients with cancer to evaluate the nutritional status. It consisted of two subscales, the patient self-assessment scale and the medical staff assessment scale. The former integrated short-term weight loss, food intake (including amount eaten, type of food, manner of eating, etc.), symptoms affecting eating, activity and physical functioning, and nutritional difficulties and activities. The latter included medical history, metabolic stress and physical examination provided by medical staff. Each item in the PG-SGA scale has a score range of 0-4. The more severe the symptoms in relation to malnutrition the higher the assigned value.

SECONDARY OUTCOMES:
nutrition-related blood indices, such as total protein (g/L), albumin (g/L), prealbumin (g/L), and hemoglobin (g/L) | T0=before the first admission to the hospital for chemotherapy, T1=2 weeks after the first chemotherapy, and T6=2 weeks after the sixth chemotherapy
  The indicators were collected from hospital electronic medical records.
inflammation-related blood indices, such as leukocytes (10^9/L), lymphocytes (10^9/L), neutrophils (10^9/L), and platelets (10^9/L) | T0=before the first admission to the hospital for chemotherapy, T1=2 weeks after the first chemotherapy, and T6=2 weeks after the sixth chemotherapy
  The indicators were collected from hospital electronic medical records.
nutrition-inflammation composite indices, such as prognostic nutritional index (PNI) and systemic immunoinflammatory index (SII) | T0=before the first admission to the hospital for chemotherapy, T1=2 weeks after the first chemotherapy, and T6=2 weeks after the sixth chemotherapy
  PNI is calculated as "albumin (g/L) + 5 × lymphocyte (10^9/L). SII is calculated as "platelet(10^9/L)×neutrophil (10^9/L)]/lymphocyte (10^9/L)

CONTACTS AND LOCATIONS:
Overall Officials: xiaojuan Tian, chief nurse, Principal Investigator — Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China